CLINICAL TRIAL: NCT04938518
Title: Investigation of the Impact of Inducible, Replication-competent Latent HIV-1 as an Impediment to HIV/AIDS Cure in the Context of Sustained Viral Suppression
Brief Title: Latent HIV-1, Viral Suppress and Hope for HIV Cure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Principal Investigator, Dr. Edward Maina, Principal Investigator, Kenya Medical Research Institute
Other Study IDs: SERU Protocol no. 3620
Record Dates: First submitted 2021-01-28; First posted 2021-06-24 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Blood will be collected from participants for plasma HIV-1 RNA, PBMCs harvesting, CD4 quantification and and cytokine analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2014, the Joint United Nations Program on HIV/AIDS (UNAIDS) issued treatment goals for Human Immunodeficiency Virus (HIV), the 90-90-90 target. It is important to track success results at each stage of the HIV continuum of care to evaluate progress towards the 90-90-90 target. Although ART can suppress HIV-1 infection to undetectable levels of plasma viremia, HIV DNA integrate and persist in resting CD4+ T cells. Most of the HIV DNA in these cells is defective and cannot cause infection. However, latent HIV-1 genomes that encode replication-competent virus can resurface once ART is discontinued. This latent reservoir is believed to be the largest impediment to a cure by ART alone. There is need for expansion of research examining HIV latency in the context of sustained viral suppression with an eye towards developing a possible cure regimen that could be used on a large scale. To date, there have been no systematic studies to quantify the latent reservoir in virally suppressed HIV-infected patients in Africa. Detecting how much of the inducible virus is left in the human body after ART poses the greatest challenge to fully curing HIV. This study is designed to enroll 222 virally suppressed HIV infected men and women, who will be prospectively followed to document antiviral cocktail, viral suppression and incidences of rebound, measure the size of the latent HIV reservoir and examine the immunological correlates of the latent reservoir. Data generated through this study will provide a clear framework for high-burden countries to reduce gaps at each stage of the HIV continuum of care, maximize linkage, retention and health outcomes.

DETAILED DESCRIPTION:
Background: Based on the 2013 Kenya AIDS Indicator Survey, 58% of people living with HIV/AIDS (PLWHA) aged 15-64 years in Kenya were eligible for Antiretroviral Therapy (ART), but only 63% of them were found to have been initiated. Previous studies have shown that an estimated 33% to 40% of patients are expected to fail treatment in the first 12 months of second-line ART. In many low and middle income countries (LMIC) with no third-line regimens available, second-line ART is the last option for patients hence failure greatly impacts patients management. A study in Kenyan national ART program suggests that about 27% of patients with second-line failure are in need of a switch to third-line therapy, with 25% demonstrating complete exhaustion of alternative first and second-line regimens. Although new drugs for HIV treatment are being developed, HIV treatment options within national programmes remain limited. Therefore, the durability of switch to second-line regimens as well as durability to second-line regimens is critical for the long-term success of ART and ultimately patient survival. Fortunately, virological (VL) failure on second-line ART does not necessarily warrant a switch to a third-line regimen, as Protease Inhibitors (PIs) have a high genetic barrier to resistance mutations, particularly among PI naïve patients. As failure on second-line ART is more related to suboptimal adherence than drug resistance, the management of VL failure on second-line typically involves intensified adherence counselling with drug substitutions recommended in cases of documented resistance mutations, severe adverse drug reactions (ADR) or drug interactions. While rates of drug substitutions and the durability of first-line ART have been previously described, there is very little information on patterns of drug substitutions for patients on second-line ART across ART national guideline-specific periods. Additionally, little is known about the impact of ART guideline changes on the durability of second-line ART and continuity of care.

While determining the durability of ART is critical in terms of monitoring success and possible ART mutations, the desired outcome is eradication of HIV by 2030.The concept of eradication of the HIV from infected patients has therefore gained much attention in the last few years. ART has changed the dynamic of the HIV epidemic through suppression of HIV-1 RNA to undetectable plasma levels. As a sign of the seriousness of countries to achieve 90-90-90, it is important to track success results at each stage of the HIV continuum of care and most importantly the viral suppression. Although antiretroviral therapy can suppress HIV-1 infection to undetectable levels of plasma viremia, HIV DNA integrate and persist in resting CD4+ T cells. Latent HIV infection of CD4+ T cells, established during the early stages of infection, necessitates lifelong ART, and treatment failure can lead to the selection of drug resistance mutations in the viral genome, which may be archived in the cellular reservoir. Most of the HIV DNA in these cells is defective and cannot cause infection. However, latent HIV-1 genomes that encode replication- competent virus can resurface once ART is discontinued. This latent reservoir having replication- competent virus has a long half-life, and is believed to be the largest impediment to a cure by ART alone. This justifies expansion of research examining HIV latency in the context of sustained viral suppression with an eye towards developing a possible cure regimen that could be used on a large scale. Recently, pharmaceutical approaches have focused on the development of molecules able to reactivate HIV from latently infected cells in order to render them susceptible to combined antiretroviral therapy (c-ART), viral cytopathic effects and host immune responses. Obviously, exposing latent virus and killing it with ART rests on an assumption that the activated virus will be susceptible to the ART a person takes. As such, it is important to discern whether reactivated HIV proviruses are susceptible to the ART regimen for maximum benefit to the patient.

The vast majority of HIV-infected individuals currently live in sub-Saharan Africa where fully suppressive ART is expanding rapidly. Due to this expansion, a large number of patients are expected to achieve full viral suppression. There is need therefore to quantify and document the size of latent HIV reservoir in virally suppressed patients in this region for individualized treatment. To date, there have been no systematic studies to quantify the latent reservoir in virally suppressed HIV-infected patients in Africa. Detecting how much of the inducible virus is left in the human body after antiretroviral therapy poses the greatest challenge to fully curing HIV. Stratifying virally suppressed patients base on the quantity of latent HIV, ART regimens and immune status may inform eligible candidates for latency reactivation care when one comes available.

Hypothesis: Archived proviruses in the latent reservoir are sustained in aviremic patients and are an impediment to HIV cure.

General Objective: Investigate the impact of inducible, replication-competent latent HIV-1 as an impediment to HIV/AIDS cure.

Objectives:

* Document treatment cocktail and determine the rate of viral rebound in aviremic patients; As a sign of the seriousness of countries to achieve 90-90-90, it is important to track success results at each stage of the HIV continuum of care. The investigator will conduct three analyses on patients: 1) Document antiviral cocktail; 2) Duration of viral suppression; 3) Monitor incidences of viral rebound. This will provide a clear framework for using data to maximize linkage, retention and health outcomes. It will also help high-burden countries to use this data at a sub-national and county level to improve service linkage and reduce gaps at each stage of the HIV continuum of care.
* Examine and measure the size of latent HIV reservoirs in virally suppressed patients; Once a patient achieves viral suppression with antiretroviral therapy, it becomes very important to tell how much virus is still left, and whether it can replicate. Such data may lead to an understanding of HIV pathogenesis and to adjust the therapy to improve the quality of life of the HIV patient and inform HIV-1 eradication strategies. This data will enable to identify patients who will be eligible candidates for cure treatment when one comes available.
* Explore the level of immune activation in virally suppressed HIV-infected patients in correlation with the size of the reservoir; In addition to harboring HIV-1 in a long-lived reservoir, individuals on ART have persistently elevated levels of inflammation and T cell activation. Abnormal inflammation and immune activation may contribute to HIV-1 persistence by driving proliferation and activation of HIV-1-infected cells and by activating uninfected cells that can support low-level viral replication. The investigator propose to evaluate sizes of HIV-1 reservoir in relation to inflammation and T cell activation in HIV-1 in aviremic patients on therapy to inform strategies aimed at reducing HIV-1 reservoirs, inflammation and activation that persist despite ART.

Study population: The study will utilize HIV-1 infected patients (18 to 70 years) attending HIV care and treatment facilities in three counties of Meru, Kilifi, and Mombasa. Analysis of medical records to document ART cocktail will be performed. Latent HIV will be determined in patients with viral suppression, defined according to WHO guideline 2016, and followed for 24 months to monitor incidences of viral rebound. A viral load threshold of <1000 copies/mL defines treatment success according to the 2016 WHO consolidated guidelines on the use of antiretroviral drugs for treating and preventing HIV infection. Hence subjects with viral load test results below the threshold will be considered as having suppressed viral loads and included in the study. Subjects with complete suppression ( with viral loads below the limit of detection) will also be included in the study.

Study sites: Participants (222) will be recruited from Tudor District Hospital in Mombasa, Malindi District Hospital in Kilifi, Maua Methodist Hospital and Meru Level Five Hospital in Meru Counties of Kenya. Sites were selected depending on volumes of HIV infected individuals registered in the HIV comprehensive care centers who have been taking HAART for at least the last 12 months and have shown virus suppression in at least one of the previous viral load test result.

Sample size calculation: Hospitals will be purposively sampled from each of the three counties of Meru, Kilifi and Mombasa due to the high HIV burden in those counties. Using the reported HIV estimated prevalence in each of the three counties, the sample size will be calculated for each county using the following formula by Armitage. Hence, sample size for;

1. Mombasa County will be; 107 HIV infected individuals
2. Meru County will be; 43 HIV infected individuals
3. Kilifi County will be; 52 HIV infected individuals

Therefore, a minimum sample size of 202 HIV infected individuals will be required for this study. However, to account for potential non-response, non-compliance, and lost to follow-up cases, 10% of the minimum sample size per county will be added hence 222 HIV infected individuals in all the three counties will be utilized.

Ethical consideration: Before commencement of the study, approval will be sought from the Centre for Microbiology Research -KEMRI, Centre Scientific Committee (CSC) as well as the KEMRI Scientific and Ethical Review Unit (SERU). Once the approval is obtained from KEMRI, The investigator will pursue approval for the study from the respective county Director of medical services where the study will be carried out. Thereafter approval from the sites (hospitals) will be sought before commencement of the study. Informed consent will be obtained from adult participants. Recruitment will be voluntary and volunteers will be encouraged to ask questions concerning their rights. Study participants who, during the course of the study are in any way incapacitated will have their consent sought afresh. Participants will not incur any costs as a result of participating in the study and will be free to withdraw from the study whenever they so wish. A coded identification number will be assigned to each participant and used only for the purposes of sample tracking. Documents linking personal identifiers and specimen results will be destroyed after the study. All information will be kept confidential.

Data collection and laboratory methods: Participant sociodemographic data, ART regimen, CD4+ cell count, opportunistic infections, World Health Organization (WHO) staging, and physician-reported adherence will be retrospectively collected from patient folders. All participants will undergo plasma HIV-1 RNA and CD4 quantification at enrollment and after every 6 months during follow up. Baseline viral load and CD4+ cell counts will be closest to ART regimen start. All HIV-1 RNA levels obtained as part of the study, will be made immediately available to the respective physician. The investigator will evaluate every paired HIV-1 viral load (VL) and CD4 count performed to analyze the durability of viral suppression and the risk of rebound among patients with virologic suppression. Time to rebound will be computed using consecutive sequences of observations for subjects whose initial two viral loads will be below the lower limit of quantification and had a viral load measurement within the duration of follow up days.

Statistical analyses: A ratio paired test or equal variance two-sample t-test will be used to calculate the significance while comparing sets of data whenever necessary. All statistical analysis will be performed using PRISM software. A P value of less or equal to 0.05 will be considered to be significant in each of the statistical analyses performed. Correlations between two independent sets of data will be performed using the Pearson correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* • HIV-1 infected patients attending HIV care and treatment facilities in three counties of Meru, Kilifi, and Mombasa.

  * Registered at the comprehensive care centre
  * Currently prescribed ART
  * Able to understand consent process
  * Have a viral load threshold of <1000 copies/mL or with viral loads below the limit of detection

Exclusion Criteria:

* • High-risk pregnancy for reasons other than HIV status (e.g., pregnancy complications, preeclampia, gestational diabetes, preterm labor)

  * Have known history of chronic diseases
  * Self-reported participation in another HIV-related study
  * Both participant and guardian unable to understand consent process
  * Planning on relocating out of study sites over the next 12 months
  * Patients of tender years(<18 yr) or extreme old age (>70 yr)
  * Incapacitated patients will not be recruited

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will utilize HIV-1 infected patients (18 to 70 years) attending HIV care and treatment facilities in three counties of Meru, Kilifi, and Mombasa. Analysis of medical records to document ART cocktail will be performed. Latent HIV will be determined in patients with viral suppression, defined according to WHO guideline 2016, and followed for 24 months to monitor incidences of viral rebound.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Types of ART regimen, and the number of aviremic patients with detectable viral loads | 12 Months
  This will entail abstracting patients' data from medical record to capture subjects' demographic data, ART regimen that the subjects had been using, viral loads measurements, duration of the ART regimen. This data will be analysed using STATA and Graphpad Prisim software to determine whether there is viral rebound in the period under study. The durability of viral suppression will be determined.
Types and Levels of Cytokines as measured by Multiplex Immunoassays | 36 Months
  Immunoassays will be carried out on blood samples from consenting patients to assess cytokine profiles. The types and levels of cytokines will be related to viral load levels and other factors. The number of aviremic patients with competent immune function will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Maina, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NASCOP, "Kenya AIDS Indicator Survey 2012:," Prelim. Rep., 2013.
- [Background] El-Khatib Z, Ekstrom AM, Ledwaba J, Mohapi L, Laher F, Karstaedt A, Charalambous S, Petzold M, Katzenstein D, Morris L. Viremia and drug resistance among HIV-1 patients on antiretroviral treatment: a cross-sectional study in Soweto, South Africa. AIDS. 2010 Jul 17;24(11):1679-87. doi: 10.1097/QAD.0b013e32833a097b. PMID 20453629
- [Background] Fox MP, Ive P, Long L, Maskew M, Sanne I. High rates of survival, immune reconstitution, and virologic suppression on second-line antiretroviral therapy in South Africa. J Acquir Immune Defic Syndr. 2010 Apr 1;53(4):500-6. doi: 10.1097/QAI.0b013e3181bcdac1. PMID 19838128
- [Background] van Zyl GU, van Mens TE, McIlleron H, Zeier M, Nachega JB, Decloedt E, Malavazzi C, Smith P, Huang Y, van der Merwe L, Gandhi M, Maartens G. Low lopinavir plasma or hair concentrations explain second-line protease inhibitor failures in a resource-limited setting. J Acquir Immune Defic Syndr. 2011 Apr;56(4):333-9. doi: 10.1097/QAI.0b013e31820dc0cc. PMID 21239995
- [Background] Dow DE, Shayo AM, Cunningham CK, Reddy EA. Durability of antiretroviral therapy and predictors of virologic failure among perinatally HIV-infected children in Tanzania: a four-year follow-up. BMC Infect Dis. 2014 Nov 7;14:567. doi: 10.1186/s12879-014-0567-3. PMID 25373425
- [Background] Inzaule SC, Hamers RL, Mukui I, Were K, Owiti P, Kwaro D, Rinke de Wit TF, Zeh C. Emergence of untreatable, multidrug-resistant HIV-1 in patients failing second-line therapy in Kenya. AIDS. 2017 Jun 19;31(10):1495-1498. doi: 10.1097/QAD.0000000000001500. PMID 28398959
- [Background] C. Orrell, "Antiretroviral adverse drug reactions and their management:," SA J CPD, vol. 26, no. 9, pp. 234-237, 2011.
- [Background] G. Meintjes, G. Maartens, A. Boulle, F. Conradie, E. Goemaere, and E. Hefer, "Adult antiretroviral therapy guideline.," South Afr J HIV Med, vol. 15, no. 4, pp. 121-143, 2014.
- [Background] Naidoo A, Naidoo K, Yende-Zuma N, Gengiah TN, Padayatchi N, Gray AL, Bamber S, Nair G, Karim SS. Changes to antiretroviral drug regimens during integrated TB-HIV treatment: results of the SAPiT trial. Antivir Ther. 2014;19(2):161-9. doi: 10.3851/IMP2701. Epub 2013 Oct 31. PMID 24176943
- [Background] Le T, Wright EJ, Smith DM, He W, Catano G, Okulicz JF, Young JA, Clark RA, Richman DD, Little SJ, Ahuja SK. Enhanced CD4+ T-cell recovery with earlier HIV-1 antiretroviral therapy. N Engl J Med. 2013 Jan 17;368(3):218-30. doi: 10.1056/NEJMoa1110187. PMID 23323898
- [Background] Dahabieh MS, Battivelli E, Verdin E. Understanding HIV latency: the road to an HIV cure. Annu Rev Med. 2015;66:407-21. doi: 10.1146/annurev-med-092112-152941. PMID 25587657
- [Background] Wensing AM, Calvez V, Gunthard HF, Johnson VA, Paredes R, Pillay D, Shafer RW, Richman DD. 2014 Update of the drug resistance mutations in HIV-1. Top Antivir Med. 2014 Jun-Jul;22(3):642-50. PMID 25101529
- [Background] PEPFAR, "Kenya Country Operational Plan," 2015.
- [Background] Inzaule S, Otieno J, Kalyango J, Nafisa L, Kabugo C, Nalusiba J, Kwaro D, Zeh C, Karamagi C. Incidence and predictors of first line antiretroviral regimen modification in western Kenya. PLoS One. 2014 Apr 2;9(4):e93106. doi: 10.1371/journal.pone.0093106. eCollection 2014. PMID 24695108
- [Background] Gandhi RT, Coombs RW, Chan ES, Bosch RJ, Zheng L, Margolis DM, Read S, Kallungal B, Chang M, Goecker EA, Wiegand A, Kearney M, Jacobson JM, D'Aquila R, Lederman MM, Mellors JW, Eron JJ; AIDS Clinical Trials Group (ACTG) A5244 Team. No effect of raltegravir intensification on viral replication markers in the blood of HIV-1-infected patients receiving antiretroviral therapy. J Acquir Immune Defic Syndr. 2012 Mar 1;59(3):229-35. doi: 10.1097/QAI.0b013e31823fd1f2. PMID 22083073
- [Background] Malnati MS, Scarlatti G, Gatto F, Salvatori F, Cassina G, Rutigliano T, Volpi R, Lusso P. A universal real-time PCR assay for the quantification of group-M HIV-1 proviral load. Nat Protoc. 2008;3(7):1240-8. doi: 10.1038/nprot.2008.108. PMID 18600229
- [Background] Cillo AR, Krishnan A, Mitsuyasu RT, McMahon DK, Li S, Rossi JJ, Zaia JA, Mellors JW. Plasma viremia and cellular HIV-1 DNA persist despite autologous hematopoietic stem cell transplantation for HIV-related lymphoma. J Acquir Immune Defic Syndr. 2013 Aug 1;63(4):438-41. doi: 10.1097/QAI.0b013e31828e6163. PMID 23493152
- [Background] Chargin A, Yin F, Song M, Subramaniam S, Knutson G, Patterson BK. Identification and characterization of HIV-1 latent viral reservoirs in peripheral blood. J Clin Microbiol. 2015 Jan;53(1):60-6. doi: 10.1128/JCM.02539-14. Epub 2014 Oct 22. PMID 25339403
- [Background] Siliciano JD, Siliciano RF. Enhanced culture assay for detection and quantitation of latently infected, resting CD4+ T-cells carrying replication-competent virus in HIV-1-infected individuals. Methods Mol Biol. 2005;304:3-15. doi: 10.1385/1-59259-907-9:003. PMID 16061962
- [Background] Biswas N, Wang T, Ding M, Tumne A, Chen Y, Wang Q, Gupta P. ADAR1 is a novel multi targeted anti-HIV-1 cellular protein. Virology. 2012 Jan 20;422(2):265-77. doi: 10.1016/j.virol.2011.10.024. Epub 2011 Nov 21. PMID 22104209
- [Background] Rosenbloom DI, Elliott O, Hill AL, Henrich TJ, Siliciano JM, Siliciano RF. Designing and Interpreting Limiting Dilution Assays: General Principles and Applications to the Latent Reservoir for Human Immunodeficiency Virus-1. Open Forum Infect Dis. 2015 Aug 26;2(4):ofv123. doi: 10.1093/ofid/ofv123. eCollection 2015 Dec. PMID 26478893
- [Background] Cillo AR, Sobolewski MD, Bosch RJ, Fyne E, Piatak M Jr, Coffin JM, Mellors JW. Quantification of HIV-1 latency reversal in resting CD4+ T cells from patients on suppressive antiretroviral therapy. Proc Natl Acad Sci U S A. 2014 May 13;111(19):7078-83. doi: 10.1073/pnas.1402873111. Epub 2014 Mar 31. PMID 24706775
- [Result] Ajose O, Mookerjee S, Mills EJ, Boulle A, Ford N. Treatment outcomes of patients on second-line antiretroviral therapy in resource-limited settings: a systematic review and meta-analysis. AIDS. 2012 May 15;26(8):929-38. doi: 10.1097/QAD.0b013e328351f5b2. PMID 22313953